CLINICAL TRIAL: NCT00502788
Title: Thalassemia Clinical Research Network - Hepatitis C Clinical Trial
Brief Title: Evaluating the Safety of Two Medications to Treat Hepatitis C in People With Thalassemia (The HepC Study)
Acronym: HepC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: National Heart, Lung, and blood Institute, National Institutes of Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 503; U01HL065238 (NIH); U01HL065238-07 (NIH)
Expanded Access: Available
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Hepatitis C; Thalassemia
MeSH Terms: conditions — Hepatitis C; Thalassemia | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Peginterferon Alfa-2a and Ribavirin — Patients will be treated with alfa-2a and ribavirin as follows:
  Peginterferon alfa-2a will be started as a dose of 180 ug subcutaneously once weekly.
  Other Names: Human recombinant E. Coli; Hoffmann-la Roche
Drug: Ribavirin — Ribavirin will be started at a dose of 800mg daily for those weighing less than or equal to 50 kg, 1000 mg daily for those with body weight 51 to 75 kg and 1200 mg daily for those with body weight > 75 kg. Ribavirin will be given orally in two divided doses. The lower dose has been included because potentially-eligible patients in the TCRN registry have a mean weight of 57 kg.

SUMMARY:
Hepatitis C is one of the most common causes of long-term liver disease in the United States. Ribavirin and peginterferon alfa-2a are two medications that are used to treat hepatitis C infection. The purpose of this study is to evaluate the safety of these two medications in adults with hepatitis C and thalassemia, a type of blood disorder.

DETAILED DESCRIPTION:
Hepatitis C is an inflammation of the liver that is caused by infection with the hepatitis C virus. Over time, people may develop liver failure, liver cancer, or cirrhosis, a condition in which the liver may become permanently scarred. Ribavirin and peginterferon alfa-2a are two medications that are used to treat hepatitis C. Ribavirin stops the hepatitis C virus from spreading inside the body, and peginterferon alfa-2a decreases the amount of hepatitis C virus in the body. Individuals with thalassemia, an inherited blood disorder that can cause anemia, often receive regular blood transfusions as part of their treatment. These individuals may have an increased risk of developing hepatitis C as a result of blood transfusions received before routine hepatitis C blood screening was available. Treating thalassemia patients with standard hepatitis C therapy can be difficult because ribavirin can worsen anemia. However, omitting ribavirin then increases the risk of hepatitis C relapse following treatment. The purpose of this study is to evaluate the safety of ribavirin and peginterferon alfa-2a for treating hepatitis C in adults with thalassemia.

This study will enroll adults with thalassemia and long-term hepatitis C. Participants will attend study visits weekly for 4 weeks, every 2 weeks until Week 24, every 4 weeks until Week 48, and then every 6 weeks until Week 72. All participants will receive a peginterferon alfa-2a injection once a week and ribavirin daily. Participants with the hepatitis C genotype 1 will receive 48 weeks of treatment; participants with all other genotypes of the disease will receive 24 weeks of treatment. A liver biopsy will occur at baseline and Week 48. The following will occur at selected study visits: physical exam, blood and urine collection, hearing and vision screening, chest x-ray, heart rate monitoring, and questionnaires to assess hepatitis C symptoms, quality of life, and depression. Participants with liver iron levels greater than 20 mg/g will undergo an echocardiogram ultrasound test every 3 months to monitor the heart.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of thalassemia
* Serum positive for hepatitis C virus RNA by polymerase chain reaction (PCR) test (using the Roche COBAS Amplicor hepatitis C virus test)
* Hepatitis B surface antigen (HBsAg) negative and HIV negative within the 12 months prior to study entry
* Liver biopsy showing histologic evidence of active hepatitis (i.e., at least grade 1 inflammation)
* Willing to use acceptable forms of contraception throughout the study

Exclusion Criteria:

* Baseline liver iron concentration greater than 40.00 mg/g dry weight (iron may be chelated and the individual re-screened). All people with liver iron levels greater than 20.00 mg/g dry weight will be permitted to enroll only if their ejection fraction is 55 or greater by echocardiography (ECHO).
* Currently participating in other interventional clinical studies
* Received interferon-alfa therapy within the 6 months prior to study entry
* Liver dysfunction, defined as international normalized ratio (INR) greater than 1.3, albumin less than or equal to 3.5g/dL, or serum bilirubin greater than 4.0 mg/dL that, in the opinion of the investigator, is not due to Gilbert's syndrome or thalassemia-related hemolysis
* Other causes of liver disease (e.g., hereditary hemochromatosis, presumed drug-associated liver disease, Wilson's disease, obesity [body mass index (BMI) greater than 30])
* Major psychiatric illness
* Neutrophil count less than or equal to 1500/mm3
* Platelet count less than or equal to 80,000/mm3
* Active alcohol abuse within the 12 months prior to study entry
* Use of illicit drugs (e.g., heroin, cocaine, angel dust) within the 2 years prior to study entry
* Alpha-fetoprotein level greater than 200 ng/mL or evidence of a liver mass lesion by either ultrasound, CT scan, or MRI scan that is suspicious for hepatocellular cancer
* Kidney insufficiency, as defined by a clinically significant abnormal serum creatinine test and confirmed by a creatinine clearance rate of less than 50 mL/min based on 24-hour urine collection. People with an elevated serum creatinine level must undergo a creatinine clearance test.
* Diabetes that, in the opinion of the investigator, is not controlled by diet, an oral hypoglycemic agent, and/or insulin
* Received an organ, limb, or bone marrow transplant
* Requires the use of certain long-term medications such as immunosuppressive medications (e.g., corticosteroids, methotrexate, azathioprine)
* Active systemic autoimmune disorder (e.g., rheumatoid arthritis, systemic lupus)
* Diagnosis or treatment of cancer within the 5 years prior to study entry, except for localized squamous or basal cell cancers treated by local excision
* Any of the following pre-existing conditions that, in the opinion of the investigator, would prevent treatment with interferon and/or ribavirin:

  1. unstable heart disease that is not controlled by medication
  2. serious cerebrovascular disease
  3. serious lung disease
* History of a seizure disorder that has not been well-controlled by anti-seizure medications within the 2 years prior to study entry
* Pregnant or breastfeeding
* Male partners of women who are pregnant
* Any other condition that, in the opinion of the investigator, would prevent study participation
* Known hypersensitivity to any study drug or their components
* Past history of multiple sclerosis, transverse myelitis, optic neuritis, papilledema, chorioretinitis, uveitis, or increased ocular pressure/glaucoma
* Currently taking hematopoietic growth factors
* Currently taking ribavirin

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2003-05; Primary Completion 2006-06 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Safety of peginterferon alfa-2a and ribavirin in individuals with thalassemia (measured by changes in liver iron stores and development of iron overload-related complications) | Measured at Week 72

SECONDARY OUTCOMES:
Mean change in hepatic iron concentration from baseline biopsy to follow-up biopsy; relationship of change to baseline level | Measured at Week 48
Transfusion frequency and volume required to maintain trough Hb 9.0-10.5 g/dL during treatment, as compared to that required in the 6 months prior to hepatitis C treatment | Measured at Week 72
Cumulate change in deferoxamine dose; evidence for deferoxamine toxicity during hepatitis C treatment | Measured at Week 72
Response rate (undetectable hepatitis C virus RNA) | Measured at Week 24 or 48
Sustained virologic response rate (undetectable hepatitis C virus RNA 24 weeks after the end of treatment) and its association with baseline hepatic iron concentration | Measured at Week 72
Rate of viral clearance from serum in the first 4 weeks of treatment, rate of early virologic response at week 12, and each rate's association with sustained virologic response | Measured at Week 72
Change in liver inflammation and fibrosis scores from baseline to 48 weeks | Measured at Week 48
Adverse events | Measured at Week 72
Cardiac adverse events, defined as either symptomatic left ventricular dysfunction requiring medication or pathologic arrhythmia requiring medication | Measured at Week 72
Quality of life | Measured at Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Jonas, MD, Study Chair — Boston Children's Hospital
Locations (5):
- United States (3):
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Weill Medical College of Cornell University, New York, New York
  - Children's Hospital Philadelphia, Philadelphia, Pennsylvania
- Toronto General Hospital, Universty Health Network, Toronto, Ontario, Canada
- University College London, London, United Kingdom